CLINICAL TRIAL: NCT06815640
Title: Effects of Intermittent Pneumatic Compression on the Recovery of High-level Cyclists
Brief Title: Effects of Intermittent Pneumatic Compression on Recovery of Cyclists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maia (Other)
Responsible Party: Principal Investigator, Filipe Silvano Pinto Maia, Principal Investigator, University of Maia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PDFM_005
Record Dates: First submitted 2025-01-12; First posted 2025-02-07 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Recovery
Keywords: sports; compression; recovery; cycling
MeSH Terms: interventions — Salvage Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IPC (Experimental): Intermittent pneumatic compression treatment (30 min peristaltic protocol, at 200mmHg)
  Interventions: Other: recovery
- Placebo (Placebo Comparator): A hydrant cream will be used as a placebo
  Interventions: Other: recovery

INTERVENTIONS:
Other: recovery — Fatigue protocol

SUMMARY:
This study aims to assess the recovery kinetics of road cyclists following a fatigue protocol (30 time trial).

ELIGIBILITY:
Inclusion Criteria:

* Road cyclists competing nationally

Exclusion Criteria:

* Injured athletes

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 21 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-07-12 (Actual)

PRIMARY OUTCOMES:
Muscle soreness | Baseline, post 30 minutes, post 24 hours, and post 48 hours
  Muscle soreness will be assessed using the likert scale of muscle soreness (ranging from 0 to 6)
Creatine Kinase | Baseline, post 30 minutes, post 24 hours, and post 48 hours
  Creatine kinase will be assessed

SECONDARY OUTCOMES:
Low frequency fatigue - Myocece Powerdex score | Baseline, post 30 minutes, post 24 hours, and post 48 hours
  Low frequency fatigue will be assessed using Myocene
4 min time trial | 24 hours post intervention
  A 4 minute time trial will be conducted at the 24th hour post-intervention.
Isometric knee extension srength | Baseline, post 30 minutes, post 24 hours, and post 48 hours
  Isometric Knee extension exercise will be assessed
Percieved fatigue | Baseline, post 30 minutes, post 24 hours, and post 48 hours
  Likert scale of percieved fatigue (ranging from 0 to 10)
Sleep questionnaires (consensus sleep diary) | Baseline, post 30 minutes, post 24 hours, and post 48 hours
  Sleep quality and quantity will be assessed using a questionnaire, based on the consensus sleep diary
Perceived recovery | Baseline, post 30 minutes, post 24 hours, and post 48 hours
  Total quality recovery scale will be used
Nutritional diaries | Baseline, post 24 hours, and post 48 hours
  Participants will be asked about their nutritional intake during the timecourse of the assessments

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade da Maia, Maia, Portugal

IPD SHARING:
Plan to Share IPD: Undecided